CLINICAL TRIAL: NCT04622293
Title: A Double-Blind, Randomized, Placebo-Controlled, Single-Center, Flexible Titration Study Evaluating the Efficacy of Solriamfetol in Treating Fatigue and Cognitive Symptoms in Adults Aged 18-65 Years With a Diagnosis of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Brief Title: A Trial of Solriamfetol in the Treatment of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rochester Center for Behavioral Medicine (Other)
Responsible Party: Principal Investigator, Joel L. Young, M.D., Medical Director, Rochester Center for Behavioral Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 102044RCT
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
Keywords: Chronic Fatigue Syndrome; Myalgic Encephalomyelitis
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Solriamfetol (Experimental): Those who are receiving solriamfetol will receive 75 mg or 150 mg. Patients will begin at a 75 mg dose and then after three days titrate up or down as needed, determined by consultation visits with primary investigator. Solriamfetol will be taken orally.
  Interventions: Drug: Solriamfetol Oral Tablet [Sunosi]
- Placebo (Placebo Comparator): Those who are not receiving solriamfetol will receive the placebo drug, which will be encapsulated in matching capsules to reduce any bias or speculation with participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol Oral Tablet [Sunosi] — Solriamfetol will be given to those participants placed in the experimental group, and given at three possible dosages ( 37.5 mg, 75 mg, and 150 mg). Solriamfetol is already FDA approved for treatment of excessive daytime sleepiness, and has been found safe to use. In this study, we are determining if solriamfetol can also be used to treat chronic fatigue syndrome.
  Other Names: Sunosi
  Arms: Solriamfetol
Drug: Placebo — A placebo encapsulated to look the same as the experimental drug will be given to the control group.
  Arms: Placebo

SUMMARY:
This study is an 8-week single center, randomized, double-blind, placebo-controlled, flexible titration trial evaluating the efficacy of solriamfetol in the treatment of fatigue symptoms in adult patients with chronic fatigue syndrome. Subjects will be randomized to a solriamfetol group or placebo group. The investigators will utilize an intent to treat model and impute data. The overall goal of this study is to determine the efficacy and effectiveness of solriamfetol for treating chronic fatigue syndrome.

DETAILED DESCRIPTION:
This will be an 8-week single center, randomized, double-blind, placebo-controlled, flexible titration trial evaluating the efficacy of solriamfetol in the treatment of fatigue symptoms in adult patients (18-65) with a diagnosis of ME/CFS. Subjects will be randomized (1:1) to a solriamfetol (flexible titration dosing) group (n=17 to 22) or placebo group (n = 17 to 22). The investigators will utilize an intent to treat model and impute data, if statistically feasible, from dropouts utilizing a MNAR (missing not at random) approach.

The trial involves primary, secondary, exploratory and safety/tolerability objectives.

Primary objective: Evaluate IMP efficacy in treating ME/CFS fatigue symptoms

Primary endpoint: Difference in means at week 8 between treatment and control groups as measured by the Fatigue Symptom Inventory.

Secondary objective: Evaluate IMP efficacy in treating ME/CFS cognitive symptoms.

Secondary endpoint: Difference in means between treatment and control groups as measured by the BRIEF-A.

Exploratory objective: Evaluate IMP efficacy in treating symptoms related to overall clinical severity/distress of patients with ME/CFS and common co-occurring conditions of ME/CFS.

Exploratory endpoints: Differences in means between treatment and control groups as measured by the Fibromyalgia Impact Questionnaire, the Sheehan Disability Scale, the Clinical Global Impression measure, and the Patient Global Impression measure.

Safety and tolerability objective: Evaluate the safety and tolerability of IMP for the treatment of patients with a diagnosis of ME/CFS.

Safety and tolerability endpoints: Frequency and severity of AEs, changes in vital signs: blood pressure, pulse rate, weight, and physical exams. Subjects will undergo a 12-lead ECG exam, Urine Drug Screens, and Urine Pregnancy Test. Suicidality will be assessed utilizing the Columbia Suicidality Severity Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must meet IOM 2015 diagnostic criteria for ME/CFS. These criteria will be assessed by obtaining clinical histories and using appropriate symptom checklists.
* All subjects must be 18-65 years of age at the time of consent.
* All sexually active males or females of child baring potential must agree to practice two different methods of birth control or remain abstinent during the course of the trial. Methods of birth control or contraception will be logged. Male and female contraception will be continued throughout the study and for 30 days after study discontinuation. Women of childbearing potential must test negative for pregnancy at the Screening Visit.
* All subjects must be able to swallow intact tablets.
* Subjects, in the opinion of the investigator, must be able to understand and comply with protocol requirements- including assessments, prescribed dosage regimens, and discontinuation of concomitant medications.
* All subjects must have a minimum level of intellectual functioning without evidence of significant general intellectual deficit, as determined by the primary investigator. Specific learning disorders will not be considered general intellectual deficits.
* All subjects must be able to provide written, personally signed and dated informed consent to participate in the study in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations before completing any study related procedures.
* All subjects must be fluent in English and have a degree of understanding sufficient to communicate suitably with the primary investigator and the study coordinator.
* Subjects must have a negative drug screen for cocaine and other illicit (illegal for recreational use in the State of Michigan) drugs excluding cannabis due to legality of cannabis in Michigan. Subjects with a positive drug screen for confirmed prescription or over the counter use of medications will require the necessary washout per PI instruction. Subjects who test positive for any prohibited medications per PI maybe permitted with PI approval. Re-tests will not be allowed for a positive screen of an illicit drug.
* All subjects must score at or above a 4 on the CGIS-S at screening.

Exclusion Criteria:

* Subjects must not be immediate family of the Investigator or others directly affiliated with the study.
* Subjects must not have received treatment with a drug that has not received regulatory approval or participated in a clinical trial within 30 days prior to screening.
* Subjects must not have medical complications arising from being severely underweight or overweight.
* Subjects must not have a current co-morbid psychiatric disorder that is uncontrolled and associated with significant symptoms or that requires a prohibited medication or behavioral modification program. Co-morbid psychiatric diagnoses will be assessed during a psychiatric intake and scoring of the MINI.
* Subjects must not currently be considered a suicide risk (as determined by the primary investigator and assessed by the C-SSRS). They must not have made a suicide attempt within the past two years. They cannot have current suicidal ideation with intent or plan to act, or current suicidal behavior.
* Subjects must not have a history of substance abuse or drug dependence according to DSM-5 criteria currently or within one year prior to study participation, excluding nicotine and caffeine. This is determined through clinical history and symptom checklist to be obtained at visit 1.
* Subjects must not test positive for an illicit substance at the time of screening.
* Subjects must not have a serious chronic or acute unstable medical condition or illness, including cardiovascular, hepatic, respiratory, or hematologic illness, narrow angle glaucoma, or other unstable medical or psychiatric conditions that in the opinion of the Investigator would compromise participation or would likely lead to hospitalization during the duration of the study. Subjects with a history of intellectual impairment or a severe learning disability are also excluded.
* Subjects must not have a history of seizure disorder (other than infantile febrile seizures), any tic disorder, current diagnosis and/or family history of Tourette's disorder.
* Subjects must not have a history of organic heart disease including coronary artery disease, past myocardial infarction, angina, arrhythmias, congestive heart failure, valvular heart disease and congenital heart disease.
* Subjects must not be likely (as assessed by the primary investigator) to add psychotropic medications, apart from their current regimen or the drug under study, to their treatment regimen during the course of the study.
* Subjects must not have been previously enrolled in this study.
* Subjects must not anticipate relocation outside the geographic range of the investigative site during participation in the study. Subjects must not have extended travel plans inconsistent with the recommended visit intervals.

Subjects must not be taking any excluded medications that cannot be discontinued prior to beginning treatment with study medication. Subjects' medical history will be reviewed by the PI and current prescription regimen will be reviewed for CNS stimulants and noradrenergic and dopaminergic medications. The PI will determine on a case by case basis if concomitant use of the patient's current prescriptions would affect response to solriamfetol and reasoning for inclusion or exclusion will be documented. Stimulant medications will be excluded (methylphenidate or amphetamine based).

* Have a known hypersensitivity, allergy intolerance or documented history of non-responsivity to NDRIs or similar medication.
* Subjects who, in the opinion of the Investigator, are unsuitable in any other way to participate in the study.
* Subjects who have taken an MAOI within 14 of the beginning of the study.
* Subjects currently taking a medication regime that would otherwise likely interfere with the efficacy of solriamfetol or the integrity of study results as determined on a case by case basis by the primary investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Symptom Inventory (FSI) | Up to 8 weeks
  This measure has excellent internal reliability and good convergent validity and construct validity. The FSI has been demonstrated to effectively discriminate between patients with clinically significant fatigue and those that do not. Its psychometric properties have repeatedly been demonstrated to support its use in research for fatigue symptoms.

SECONDARY OUTCOMES:
BRIEF-A | Up to 8 weeks
  The BRIEF-A is a comprehensive measure of executive functioning, examining 8 cognitive tasks. It is non-diagnosis specific and applicable for use with a variety of cognition-impacting conditions

OTHER OUTCOMES:
Clinical Global Impression (CGI-I and CGI-S) | Up to 8 weeks
  The CGI-S measures severity at baseline and the CGI-I measures improvement. It is commonly utilized across FDA-regulated trials. The Patient Global Impression (PGI-I and PGI-S) measure was created to tack efficacy in studies involving incontinence, and has become widely used in clinical research to capture change in functioning from the perspective of the patient.
Young CFS Scale | Up to 8 weeks
  Due to the strong research and clinical need for a better self-report diagnostic screening tool for ME/CFS that can also reflect changes in symptoms due to treatment, this trial will assist in the development of a proposed measure of ME/CFS, entitled the "Young CFS Scale." Part of the validation of this measure will be analysis of its relationship with other measures in measuring ME/CFS in clinical samples.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Young, MD, Principal Investigator — Rochester Center for Behavioral Medicine
Locations (1):
- Rochester Center for Behavioral Medicine, Rochester Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data that was collected during this study.

REFERENCES:
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Donovan KA, Jacobsen PB, Small BJ, Munster PN, Andrykowski MA. Identifying clinically meaningful fatigue with the Fatigue Symptom Inventory. J Pain Symptom Manage. 2008 Nov;36(5):480-7. doi: 10.1016/j.jpainsymman.2007.11.013. Epub 2008 May 20. PMID 18495413
- [Background] Donovan KA, Jacobsen PB. The Fatigue Symptom Inventory: a systematic review of its psychometric properties. Support Care Cancer. 2010 Feb;19(2):169-85. doi: 10.1007/s00520-010-0989-4. Epub 2010 Sep 8. PMID 20824482
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Strollo PJ Jr, Hedner J, Collop N, Lorch DG Jr, Chen D, Carter LP, Lu Y, Lee L, Black J, Pepin JL, Redline S; Tones 4 Study Investigators. Solriamfetol for the Treatment of Excessive Sleepiness in OSA: A Placebo-Controlled Randomized Withdrawal Study. Chest. 2019 Feb;155(2):364-374. doi: 10.1016/j.chest.2018.11.005. Epub 2018 Nov 22. PMID 30471270
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Derived] Young JL, Powell RN, Powell A, Welling LLM, Granata L, Saal J. Solriamfetol improves daily fatigue symptoms in adults with myalgic encephalomyelitis/chronic fatigue syndrome after 8 weeks of treatment. J Psychopharmacol. 2025 Nov;39(11):1268-1276. doi: 10.1177/02698811251368371. Epub 2025 Sep 16. PMID 40958377